CLINICAL TRIAL: NCT01987947
Title: A Study of Quilizumab Versus Placebo in Patients With Refractory Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GX29107
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Urticaria
Keywords: MEMP1972A
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Quilizumab (Active Comparator)
  Interventions: Drug: Quilizumab

INTERVENTIONS:
Drug: Placebo — Two administrations by subcutaneous injection
  Arms: Placebo
Drug: Quilizumab — Two administrations by subcutaneous injection
  Arms: Quilizumab

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled, parallel-group study will assess the efficacy and safety of additional quilizumab therapy in adult patients with Chronic Spontaneous Urticaria resistant to antihistamine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CSU refractory to H1 antihistamines with/without LTRAs, as defined by the following:
* The presence of itch and hives for > 6 consecutive weeks at any time prior to enrollment despite use of H1 antihistamines during this time period
* UAS7 score greater than 16 and itch component of UAS7 greater than 8 during 7 days prior to Day 1. Patients must have been on daily stable doses of H1 antihistamine for at least 3 consecutive days immediately prior to the screening visit and must document current use at screening
* CSU diagnosed for more than 6 months
* Patients must have a minimum diary compliance (6 out of 7 consecutive days) prior to Day 1

Exclusion Criteria:

* Treatment with an investigational agent within 30 days of screening, and previous treatment with monoclonal antibody therapies used to treat CSU 9 months prior to screening
* Chronic urticarias other than CSU, including the following: Acute, solar, cholinergic, heat, cold, aquagenic, delayed pressure or contact.
* Other diseases and conditions with symptoms of urticaria.
* Routine doses of the following medications within 30 days prior to screening: systemic or topical corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide
* IV immunoglobulin G (IVIG), or plasmapheresis within 30 days prior to screening
* Patients with cancer, history of cancer considered uncured or in complete remission for < 10 years, or currently under work-up for suspected cancer except non-melanoma skin cancer that has been treated or excised and is considered resolved
* History of anaphylactic shock without clearly identifiable avoidable antigen
* Presence of clinically significant cardiovascular, neurological, psychiatric, metabolic or other pathological conditions.
* Medical examination or laboratory findings that suggest the possibility of decompensation of co-existing conditions for the duration of the study.
* Evidence of current drug or alcohol abuse
* Nursing women and women of childbearing potential, unless using effective contraception as defined by protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: Absolute change from baseline to Week 20 in the weekly itch score. | 21 weeks
Safety: Incidence & severity of adverse events. | Approximately 30 weeks
Safety: Incidence of anti-therapeutic antibodies. | Approximately 30 weeks

SECONDARY OUTCOMES:
Efficacy: Absolute change from baseline to Week 4 in the weekly itch score. | 5 weeks
Efficacy: Absolute change from baseline to Week 20 in the UAS7 aggregate score. | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (3):
- Toronto, Ontario, Canada
- Germany (2):
  - Berlin
  - Mainz